CLINICAL TRIAL: NCT00725751
Title: Evaluation of Treatment of Chronic Hepatitis C With Pegylated Interferon and Ribavirin in Patients With/Without Substitution Therapy in Austria
Brief Title: Treatment of Chronic Hepatitis C With Pegylated Interferon and Ribavirin in Participants With/Without Substitution Therapy (P05255)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P05255
Record Dates: First submitted 2008-07-25; First posted 2008-07-30 (Estimated); Results first posted 2012-04-23 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PegIFN-2b/ribavirin with substitution therapy: Participants in this cohort received antiviral treatment and substitution therapy (opioid medicines with long-lasting effects [methadone + buprenorphine] or morphine)
  Interventions: Biological: Pegylated interferon alfa-2b (PegIFN-2b); Drug: Ribavirin
- PegIFN-2b/ribavirin without substitution therapy: Participants in this cohort received antiviral treatment but did not receive substitution therapy (opioid medicines with long-lasting effects [methadone + buprenorphine] or morphine)
  Interventions: Biological: Pegylated interferon alfa-2b (PegIFN-2b); Drug: Ribavirin

INTERVENTIONS:
Biological: Pegylated interferon alfa-2b (PegIFN-2b) — PegIFN-2b administered according to European labeling.
  Other Names: PegIntron; SCH 54031
Drug: Ribavirin — Ribavirin administered according to European labeling.
  Other Names: Rebetol; SCH 18908

SUMMARY:
Although injection drug users represent the majority of new and existing cases of infection with hepatitis C virus (HCV), many lack access to treatment because of concerns about adherence, effectiveness, and reinfection. On the basis of a small but growing body of evidence showing that injection drug users can undergo treatment for HCV infection successfully, the 2002 NIH Consensus Statement on Hepatitis C has recommended that substance users be treated for HCV infection on a case-by-case basis. In this study, all patients will receive pegylated interferon alfa-2b (PegIFN-2b) and ribavirin according to European labeling; one cohort of participants will also be receiving substitution therapy (opioid medicines with long-lasting effects [methadone + buprenorphine] or morphine).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with hepatitis C

Exclusion Criteria:

* According to the products' European labeling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients receiving treatment for hepatitis C with/without substitution therapy at sites in Austria.
Sampling Method: Non-Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2007-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 353 participants were enrolled on the study; 348 were treated.
Groups:
- PegIFN-2b/Ribavirin With Substitution Therapy: Participants in this group received antiviral treatment and substitution therapy (opioid medicines with long-lasting effects [methadone + buprenorphine] or morphine)
- PegIFN-2b/Ribavirin Without Substitution Therapy: Participants in this group received antiviral treatment but did not receive substitution therapy (opioid medicines with long-lasting effects [methadone + buprenorphine] or morphine)
Period: Overall Study
Arm/Group | PegIFN-2b/Ribavirin With Substitution Therapy | PegIFN-2b/Ribavirin Without Substitution Therapy
Started | 90 | 258
Completed | 56 | 150
Not Completed | 34 | 108

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PegIFN-2b/Ribavirin With Substitution Therapy | PegIFN-2b/Ribavirin Without Substitution Therapy | Total
Number analyzed (Participants) | 90 | 258 | 348
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.38 (9.51) | 42.26 (12.62) | 39.71 (12.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 96 | 125
  Male | 61 | 162 | 223
Region of Enrollment [Number; unit: participants]
  Austria | 90 | 258 | 348

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed Treatment With PegIFN-2b/Ribavirin
Description: For participants with Genotype 1 or 4 completion of treatment was at Week 48; for participants with Genotype 2, 3, or 1 with low viral load or rapid virologic response, completion of therapy was at Week 24.
Time Frame: 24 to 48 weeks
Population: Participants who received at least one dose of PegIFN-2b/ribavirin
Measure: Number; unit: participants
Arm/Group | PegIFN-2b/Ribavirin With Substitution Therapy | PegIFN-2b/Ribavirin Without Substitution Therapy
Number analyzed (Participants) | 90 | 258
participants | 56 | 150

2. Secondary Outcome: Number of Participants Who Achieved Sustained Virologic Response (SVR)
Description: SVR was defined as a hepatitis C virus (HCV) ribonucleic acid (RNA) value below the limit of detection by polymerase chain reaction (PCR) analysis. For participants with Genotype 1 or 4 completion of treatment was at Week 48; for participants with Genotype 2, 3, or 1 with low viral load or rapid virologic response, completion of therapy was at Week 24.
Time Frame: 24 weeks after the end of treatment (i.e. 48 or 72 weeks depending on genotype)
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | PegIFN-2b/Ribavirin With Substitution Therapy | PegIFN-2b/Ribavirin Without Substitution Therapy
Number analyzed (Participants) | 90 | 258
participants | 42 | 111

3. Secondary Outcome: Number of Participants Who Received Antiviral Treatment Who Were Also on Substitution Therapy
Description: This measure was the number of all of the participants who received antiviral treatment who also received substitution therapy.
Time Frame: Day 1
Population: Participants who received at least one dose of antiviral treatment.
Measure: Number; unit: participants
Groups:
- All Participants: Participants who received at least one dose of antiviral treatment and substitution therapy (opioid medicines with long-lasting effects [methadone + buprenorphine] or morphine)
  Participants who received at least one dose of antiviral treatment and did not receive substitution therapy (opioid medicines with long-lasting effects [methadone + buprenorphine] or morphine)
Arm/Group | All Participants
Number analyzed (Participants) | 348
participants | 90

ADVERSE EVENTS:
Description: All participants who received at least one dose of study therapy.
Arm/Group | PegIFN-2b/Ribavirin With Substitution Therapy | PegIFN-2b/Ribavirin Without Substitution Therapy
Serious Adverse Events (participants affected / at risk) | 1/90 | 10/258
Other Adverse Events (participants affected / at risk) | 18/90 | 35/258
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegIFN-2b/Ribavirin With Substitution Therapy (N=90) | PegIFN-2b/Ribavirin Without Substitution Therapy (N=258)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Accidental death (General disorders) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegIFN-2b/Ribavirin With Substitution Therapy (N=90) | PegIFN-2b/Ribavirin Without Substitution Therapy (N=258)
Fatigue (General disorders) | 8 (8) | 12 (12)
Influenza like illness (General disorders) | 10 (10) | 14 (15)
Weight decreased (Investigations) | 5 (5) | 6 (6)
Headache (Nervous system disorders) | 5 (5) | 5 (5)
Depression (Psychiatric disorders) | 5 (5) | 7 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No